CLINICAL TRIAL: NCT05794321
Title: Investigating the Use of Intravenous Tranexamic Acid in Gender Affirming Mastectomy
Acronym: IVTXA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Esther Kim, MD, Associate Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-38580
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Hematoma; Postoperative Seroma
Keywords: Gender Affirming Mastectomy; Tranexamic Acid; IV TXA

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to treatment arms. One treatment arm will include the use of IV TXA, the other treatment arm will receive the standard of care for treatment. Patients then remain in that same treatment arm throughout the course of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IV TXA Group (Experimental): Patients in the experimental group will receive a loading dose of IV tranexamic acid (TXA) at a concentration of 1g/10ml over a period of 10 minutes, administered immediately following anesthesia induction. Postoperative care will be standard and based on established UCSF guidelines.
  Interventions: Drug: Intravenous TXA
- Control Group (No Intervention): Patients in the control group will not receive any IV TXA intraoperatively and will undergo a traditional gender affirming mastectomy following the established standard of care.

INTERVENTIONS:
Drug: Intravenous TXA — Patients in the experimental group will receive a loading dose of tranexamic acid (TXA) at a concentration of 1g/10ml over a period of 10 minutes, administered immediately following anesthesia induction.
  Arms: IV TXA Group

SUMMARY:
Gender affirming surgeries (GAS) have been steadily increasing in the US, with the gender affirming mastectomy (GAM) being the most common surgery performed. Complications associated with these surgeries include hematoma and seroma. Prior studies in orthopedics, plastic surgery, and trauma have shown significant reduction of bleeding and ecchymosis with the use of tranexamic acid (TXA). TXA is a synthetic amino acid that blocks plasminogen conversion to plasmin, to stabilize clot formation. The intravenous (IV) efficacy in reducing hematoma rates has been established in implant-based breast reconstruction, as well as in reduction mammaplasty. However, there are currently no studies investigating the use of IV TXA in patients undergoing GAM.

The investigators propose a single-center, prospective randomized control trial to evaluate the efficacy and safety of intravenous tranexamic acid in decreasing hematoma and seroma rates for top surgery patients at UCSF. Patients will be randomized into two groups, an experimental group receiving IV TXA and a control group that will not receive IV TXA.

Patients in the experimental group will receive a loading dose of tranexamic acid (TXA) at a concentration of 1g/10ml over a period of 10 minutes, administered immediately following anesthesia induction. Patients will be excluded if they have a history of coagulopathy, bleeding disorders or prior chest surgery. Demographic data, surgical characteristics, and postoperative outcomes will also be recorded and analyzed. The investigators hypothesize that the use of IV TXA will significantly reduce hematoma, seroma, postoperative drain output, and time to drain removal in patients undergoing GAM.

Aim 1: To evaluate the effectiveness of IV TXA in reducing intraoperative bleeding, post-operative hematoma and seroma formation, drain output, and time to drain removal in patients undergoing GAM.

Aim 2: To compare the incidence of thromboembolic events and wound complications between patients receiving IV TXA and those who do not after GAM.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled single-surgeon trial performed at the University of California San Francisco that investigates the use of IV TXA in patients undergoing GAM. All patients who meet WPATH guidelines for GAM, undergo GAM, ASA I-III, and are >18 years old will have the opportunity to be enrolled. Patients will be randomized by a random computer generator and will be notified after randomization as to which group they are assigned.

The investigators will enroll patients into this prospective trial investigating the effect of IV TXA on postoperative bleeding, hematoma, seroma, drain output, and time to drain removal. Patients will be randomized into two groups, an experimental group receiving IV TXA and a control group that will not receive IV TXA. Patients will be excluded if they are <18 years old, have a history of prior chest surgeries, coagulopathy or bleeding disorders, and have a history of thromboembolic events including deep vein thrombosis or pulmonary embolism. Patients will also be excluded if they are chronically anticoagulated, are on antiplatelet medications or have ever had an adverse reaction to IV TXA.

All patients who are being scheduled to undergo bilateral mastectomy with immediate reconstruction will be recruited to participate in the study. Patients will be consented to participate in the preoperative visit.

Experimental Group: Patients in the experimental group will receive a loading dose of tranexamic acid (TXA) at a concentration of 1g/10ml over a period of 10 minutes, administered immediately following anesthesia induction. Postoperative care will be standard and based on established UCSF guidelines.

Control Group: Patients in the control group will not receive any TXA intraoperatively and will undergo a traditional GAM.

Tranexamic Acid is available as a sterile, single-dose. This 1g vial is readily available in the anesthesia cart in the operating room. Immediately following induction, the anesthesia team will administer 1g of TXA intravenously. After obtaining hemostasis and irrigating as per standard practice, anesthesia shall not use any other hemostatic agents.

Post-procedure, each patient will be provided with standard postoperative instructions which will include a chart to record daily drain outputs for the right and left sides. At subsequent postoperative visits, drain output will be assessed at each clinic visit to determine timing for removal. The total drain output will be measured by the patient and later logged into our chart for later analysis. Drains will be removed per standard practice at our institution which is when they have produced < 30cc/day for at least 3 days.

At each clinic visit, the investigators will assess for clinical signs of hematoma and seroma, and objectively measure aggregate drain output. Demographic data, surgical characteristics, and postoperative outcomes such as hematoma, seroma, drain output, wound complications, surgical site infections, and thromboembolic events will be recorded and analyzed. These outcomes will be evaluated in the immediate 3-month postoperative period, with a 1-year follow-up review of patient charts. The primary outcomes will include the presence of hematoma, seroma, and drain output, and time to drain removal, while the secondary outcomes will consist of thromboembolic events and wound complications.

Patients will be managed for hematoma and seroma as per standard procedure, whether with ultrasound, clinic aspiration, IR drain placement, or return to the operating room as deemed necessary by the senior surgeon.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age
2. All patients who undergo gender affirming mastectomy at UCSF
3. ASA I-III,
4. Ability to understand a written informed consent document, and the willingness to sign it.
5. Patients who fulfil WPATH guidelines/criteria for undergoing GAM. WPATH Criteria include: Persistent, well-documented gender dysphoria; capacity to make a fully informed decision and to consent for treatment; age of majority in a given country; if significant medical or mental health concerns are present, they must be reasonably well controlled; 12 continuous months of hormone therapy as appropriate to the patient's gender goals (for two referrals by a mental health professional).

Exclusion Criteria:

1. <18 years old
2. Unable to consent for themselves
3. History of coagulopathy or bleeding disorders
4. History of thromboembolic events including deep vein thrombosis or pulmonary embolism.
5. Patients who are chronically anticoagulated, are on antiplatelet medications or have ever had an adverse reaction to IV TXA.
6. Prior history of chest surgery.
7. Known hypersensitivity or allergy to TXA
8. Patients with severe renal impairment .

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Clinically Significant Hematomas | Up to 3 months
  Hematoma will be defined as a collection of blood outside of blood vessels that requires intervention such as aspiration or surgical drainage. Hematomas that are smaller or that resolve without intervention will not be included in the analysis. All patients will undergo a physical examination during their postoperative clinic visits to assess for hematoma formation. Patients who develop symptoms of hematoma after discharge will be instructed to seek medical attention immediately. Hematoma will be assessed immediately after mastectomy, and then at their one week postoperative clinic visit. Patients will also be instructed to report any symptoms of hematoma to their healthcare provider after discharge. Data on hematoma will be collected as a binary outcome (yes/no), as well as the size of the hematoma and type of intervention. Statistical analysis will be used to determine the factors associated with hematoma development after mastectomy.
Number of Participants with Clinically Significant Seromas | Up to 3 months
  Seroma will be defined as a collection of fluid that accumulates in the surgical site after mastectomy that requires intervention such as aspiration or surgical drainage. Seromas that are smaller or that resolve without intervention will not be included in the analysis. All patients will undergo a physical examination during their postoperative clinic visits to assess for seroma formation. Seroma will be assessed immediately after mastectomy, and then at their one postoperative clinic visit. Patients will also be instructed to report any symptoms of seroma to their healthcare provider after discharge. Data on seroma will be collected as a binary outcome (yes/no), as well as the type of intervention, and the duration of symptoms. Statistical analysis will be used to determine the factors associated with seroma development after mastectomy.
Total Patient Drain Output | Up to 3 months
  Drain output will be defined as the amount of fluid (in milliliters) collected in surgical drains after mastectomy. The volume of fluid collected will be recorded by patients daily until the drains are removed. All patients will have surgical drains placed after mastectomy. Patients will be instructed to report any unusual drainage or bleeding to their healthcare provider. Data on drain output will be collected as a continuous variable, as well as the duration of drain placement. Statistical analysis will be used to determine the factors associated with increased drain output after mastectomy.
Time to Drain Removal | Up to 3 months
  Time to drain removal will be defined as the number of days from mastectomy surgery to the day the surgical drains are removed. The timing of drain removal will be determined by the primary surgeon, based on the amount and character of fluid collected in the drain, and the presence of factors such as infection, hematoma, or seroma. However, drains will typically be removed when they have produced < 30cc/day for at least 3 days. The timing of drain removal will be recorded by nursing staff at the time of removal. Data on time to drain removal will be collected as a continuous variable, as well as the reason for early or delayed drain removal. Statistical analysis will be used to determine the factors associated with longer time to drain removal after mastectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Kim, MD, Principal Investigator — UCSF Department of Plastic & Reconstructive Surgery
Locations (1):
- UCSF Department of Plastic & Reconstructive Surgery, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Only researchers designated on the IRB study application will be allowed to access patient data.

REFERENCES:
- See also: Gender-Affirming Mastectomy in Transmasculine Patients — https://journals-lww-com.ucsf.idm.oclc.org/annalsplasticsurgery/Fulltext/2021/07000/Gender_Affirming_Mastectomy_in_Transmasculine.5.aspx
- See also: Topical moistening of mastectomy wounds with diluted tranexamic acid to reduce bleeding: randomized clinical trial — https://pubmed-ncbi-nlm-nih-gov.ucsf.idm.oclc.org/32207575/
- See also: Early Postoperative Outcomes of Breast Cancer Surgery in a Developing Country — https://www.cureus.com/articles/39967-early-postoperative-outcomes-of-breast-cancer-surgery-in-a-developing-country#!/
- See also: The Use of Hemostatic Agents to Decrease Bleeding Complications in Breast Cancer Surgery — https://journals-sagepub-com.ucsf.idm.oclc.org/doi/full/10.1177/00031348211029866
- See also: U.S. Sex Reassignment Surgery Market Size, Share & Trends Analysis Report by Gender Transition (Male To Female, Female To Male), and Segment Forecasts, 2022-2030 — https://www.researchandmarkets.com/reports/5649369/u-s-sex-reassignment-surgery-market-size-share
- See also: Efficacy of Tranexamic Acid in Reducing Seroma and Hematoma Formation Following Reduction Mammaplasty — https://pubmed-ncbi-nlm-nih-gov.ucsf.idm.oclc.org/35029651/
- See also: The Usage of Intravenous Tranexamic Acid in Reduction Mammaplasty Safely Reduces Hematoma Rates — https://pubmed-ncbi-nlm-nih-gov.ucsf.idm.oclc.org/36729851/
- See also: Intravenous Tranexamic Acid in Implant-Based Breast Reconstruction Safely Reduces Hematoma without Thromboembolic Events — https://pubmed-ncbi-nlm-nih-gov.ucsf.idm.oclc.org/32740567/
- See also: Tranexamic Acid general StatPearls — https://www.ncbi.nlm.nih.gov/books/NBK532909/